CLINICAL TRIAL: NCT04658615
Title: Effects of Non-surgical Periodontal Therapy (NSPT) in Patients With and Without Rheumatoid Arthritis (RA)
Brief Title: Periodontal Treatment in Rheumatoid Arthritis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-2016
Record Dates: First submitted 2020-11-23; First posted 2020-12-08 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Rheumatoid Arthritis; Periodontitis
MeSH Terms: conditions — Arthritis, Rheumatoid; Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group with rheumatoid arthritis (Other): Non-surgical periodontal therapy (NSPT)
  Interventions: Procedure: Non-surgical periodontal therapy
- group without rheumatoid arthritis (Other): Non-surgical periodontal therapy (NSPT)
  Interventions: Procedure: Non-surgical periodontal therapy

INTERVENTIONS:
Procedure: Non-surgical periodontal therapy — A single 1-hour session of full-mouth debridement with an ultrasonic device under local anesthesia

SUMMARY:
Periodontitis is a chronic disease that leads to the loss of teeth. It has been associated to rheumatoid arthritis (RA). Periodontal therapy (NSPT) has been shown to have systemic effects. The objective of this study was to compare the effects of non-surgical periodontal therapy on biochemical parameters of rheumatoid arthritis (RA), periodontal parameters and quality of life in patients with and without RA.

Adult patients with and RA and periodontitis can participate in the study. Participants benefit from the effects of conventional tooth cleaning (periodontal therapy) and oral hygiene instructions. There are no significant risk associated with periodontal therapy.

The study is conducted at the Universidad de Antioquia in Medellin, Colombia. The study is set to start 2019 and end mid 2021. The study is funded by a grant from the Universidad de Antioquia. Contact person: Javier Enrique Botero (javier.botero@udea.edu.co)

DETAILED DESCRIPTION:
After participants are screened for inclusion, serum samples will be collected for the analysis of C-reactive protein (CRP; mg/L), rheumatoid factor (RF; UI/mL) and anti-citrullinated protein antibodies (ACPAs; UI/mL) in a reference laboratory. A complete periodontal chart will be carried out at six sites per tooth excluding third molars by a single experienced clinician using a calibrated probe (Hu-Friedy Mfg. Co.). Subgingival plaque samples will be collected by means of paper points inserted to the bottom of the pocket and processed immediately for culture analysis and detection of Porphyromonas gingivalis. RA patients will be examined by an experienced rheumatologist to determine their Disease Activity Score (DAS-28). All examinations will be taken at baseline and repeated 3 months after intervention.

Non-surgical periodontal therapy (NSPT) will be administered on the following 5 days of inclusion. A single 1-hour session of full-mouth debridement with an ultrasonic device will be carried out in each participant under local anesthesia by an experienced clinician. After NSPT is completed, each patient will receive oral hygiene instructions and oral care pack including toothbrush and toothpaste (toothbrush Vitis Encias Medium; Toothpaste Vitis Encias; Dentaid, Colombia).

Demographic ,clinical history as well as medication data for all participants will be collected. Periodontal parameters of PD (mm), PAL (mm) and BOP (%) will be recorded at each visit. The stage and grade of periodontitis will be established according to the new classification of periodontal diseases (Papapanou et al. 2018). The clinician who records data will not be blinded to the condition of the patients.

Sample size was calculated to detect a 50 % change in CRP with a power of >80% (alpha 0,05) which resulted in 15 per group (Cosgarea et al. 2018). Considering possible dropouts, 20 participants will be included per group. Randomization will not be performed since the purpose was to compare the effects of NSPT in patients with and without RA. The clinical investigator who records periodontal parameters will be calibrated for repeated measurements before patient inclusion (Kappa value was ≥0.80 for PAL and PD). Continuous variables will be presented as the mean and 95% confidence interval (CI) or median [interquartile range] when appropriate. Change in biochemical markers (CRP, RF, ACPAs) and periodontal parameters (PAL, PD, BOP, microbial counts) will be expressed as the delta (∆) from baseline to 3 months after intervention. Differences in means will be determined by the student t test for paired and unpaired samples or non-parametric tests when appropriate. Categorical variables will be presented as frequencies (%) and analyzed in contingency tables and X2. Logistic regression analysis for categorical variables and linear models will be used to test for associations and the odds ratio with 95%CI will be calculated. The primary analysis will be performed as intention to treat and then compared to per-protocol analysis results. The level of statistical significance will be set at 5% (P≤0,05).

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years old; diagnosis of RA according to the American College of Rheumatology with DAS-28 score ≥ 3.2 and no change in RA medication in the previous 3 months;
* at least 15 teeth excluding third molars;
* ≥2 non-adjacent teeth interproximal sites with loss of periodontal attachment level (PAL) ≥ 2 mm; or buccal or oral PAL ≥3 mm with pocketing >3 mm is detectable at ≥2 teeth.
* Patients without RA met the same criteria except for the diagnosis of RA.

Exclusion Criteria:

* periodontal treatment or use of antibiotics in the previous 3 months.
* diabetes, liver disease, head and neck radiation therapy.
* pregnancy
* HIV
* use of cyclosporine.
* Smoking, use of hypertension and hyperlipidemia medication were not exclusion criteria and were recorded accordingly.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in C reactive protein | 3 months
  change in C-reactive protein levels (mg/L) measured as the difference between the baseline and 3-month examination.

SECONDARY OUTCOMES:
Change in rheumatoid factor (RF) | 3 months
  change in RF levels (UI/mL) measured as the difference between the baseline and 3-month examination.
Change in anti-citrullinated protein antibodies (ACPAs) | 3 months
  change in ACPA levels (UI/mL) measured as the difference between the baseline and 3-month examination
Change in periodontal attachment level (PAL) | 3 months
  change in PAL (mm) measured as the difference between the baseline and 3-month examination
Change in probing depth (PD) | 3 months
  change in PD (mm) measured as the difference between the baseline and 3-month examination
Change in bleeding on probing (BOP) | 3 months
  change in BOP (%) measured as the difference between the baseline and 3-month examination
Change in microbial counts | 3 months
  change in subgingival microbial counts (% total colony counts) measured as the difference between the baseline and 3-month examination
Change in quality of life | 3 months
  Change in The Short Form ( SF36) Health Survey measured as the difference between the baseline and 3-month examination. It is converted to a 0-100 scale.The lower the score the more disability. The higher the score the less disability.
Change in oral health profile | 3 months
  Change in Oral Health Impact Profile (OHIP-14) measured as the difference between the baseline and 3-month examination. The OHIP-14 scores can range from 0 to 56 and are calculated by summing the ordinal values for the 14 items. Higher scores indicate worse and lower scores indicate better oral health quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Javier E Botero, PhD, Principal Investigator — Universidad de Antioquia
Locations (1):
- Facultad de Odontologia, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: Yes
Raw data will be available at the end of the study upon request
Supporting Information: Study Protocol, SAP
Time Frame: june 2021 to june 2022
Access Criteria: For secondary analyses upon request and giving full credits and participation

REFERENCES:
- [Derived] Botero JE, Posada-Lopez A, Mejia-Vallejo J, Pineda-Tamayo RA, Bedoya-Giraldo E. Effects of nonsurgical periodontal therapy in patients with rheumatoid arthritis: a prospective before and after study. Colomb Med (Cali). 2021 Sep 30;52(3):e2095051. doi: 10.25100/cm.v52i3.5051. eCollection 2021 Jul-Sep. PMID 35431355